CLINICAL TRIAL: NCT05270915
Title: Testing a Family Supportive End of Life Care Intervention in a Chinese Neonatal Intensive Care Unit: A Quasi-experimental Study With a Non-randomized Controlled Trial Design
Brief Title: End of Life Care in Neonatal Intensive Unite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HN08
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Palliative Care
Keywords: neonatal death; end-of-life care; infants; parents; neonatal intensive care; family-centered care
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family supportive EOLC (Experimental): The intervention 'family supportive EOLC' was developed based on the international guidelines of family-centered care (25) with additional aspects of care and support. The investigators designed a separated single-bedded EOLC room for the infant and parents. Other family members, such as grandparents or siblings, were allowed to visit the infant and parents. The design of the room included the option for parents to stay comfortably on a sofa to relax and to play soothing music. Parents were encouraged to stay as long as they want and participate in basic care including physical contact with their infant. The nurses supported the parents in creating commemorative items such as a 'Yuan man' box with photos, baby handprint cards, footprint cards, a lock of hair and other precious memory items. A psychologist, in collaboration with our NICU, and a neonatologist supported the parents by individual interviews.
  Interventions: Behavioral: Family supportive care in EOLC
- The standard EOLC (Active Comparator): The standard EOLC included the international guidance of palliative care and EOLC in neonatology (21-23). In China, parents are often the decision-makers of their infant's treatment and the NICU clinicians usually respect the parent's decision (24). After parents have decided to withdraw treatment, standard EOLC is initiated and includes monitoring of vital signs and withholding or withdrawing rescue procedures such as intubation and intravenous infusion. Unnecessary lines are removed and pain management is provided by analgesia. Comfort care is provided by nurses including basic care such as skin care and oral care. After the infant died, the NICU physician informs the parents by phone.
  Interventions: Behavioral: Family supportive care in EOLC

INTERVENTIONS:
Behavioral: Family supportive care in EOLC — The investigators designed a separated single-bedded EOLC room for the infant and parents. Other family members, such as grandparents or siblings, were allowed to visit the infant and parents. The design of the room included the option for parents to stay comfortably on a sofa to relax and to play soothing music. Parents were encouraged to stay as long as they want and participate in basic care including physical contact with their infant. The nurses supported the parents in creating commemorative items such as a 'Yuan man' box with photos, baby handprint cards, footprint cards, a lock of hair and other precious memory items. A psychologist, in collaboration with our NICU, and a neonatologist supported the parents by individual interviews.

SUMMARY:
In China, neonatal death on 2019 was 3.5 per 1000 live births, which counts around 57,000 deaths. In mainland China, parents are mostly the main decision-makers in withdrawing life-sustaining treatments in infants and neonatologists often follow the wishes of the parents. However, there is limited experience in supporting parents after the decision is made to withdraw treatment. The aim of this study was to develop and test a family supportive end-of-life care intervention to decrease parental depression and increase parent satisfaction. Investigators indicated that providing a comfortable environment and supportive care to parents during the final days of life of an infant decrease their depression and increases parent satisfaction. The NICUs in mainland China and beyond might consider involving parents in end-of-life care by providing a single room, have a dedicated psychologist available and provide supportive commemoration materials.

DETAILED DESCRIPTION:
Neonatal death often occurs in tertiary Neonatal Intensive Care Units (NICUs). In China, end-of-life-care (EOLC) does not always involve parents. The aim of this study is to evaluate a parent support intervention to integrate parents at the end of life of their infant in the NICU.

A quasi-experimental study using a non-randomized clinical trial design was conducted between May 2020 and September 2021. Participants were infants in an EOLC pathway in the NICU and their parents. Parents were allocated into a family supportive EOLC intervention group or a standard EOLC group based on their wishes. Primary outcomes were depression (Edinburgh Postnatal Depression Scale for mothers; Hamilton Depression rating scale for fathers) and satisfaction. Student t-test for continuous variables and the Chi-square test categorical variables were used in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infants whose treatment was withdrawn at Corrected Gestational Age (CGA) less than 28 days and their parents.

Exclusion Criteria:

* Infants with an expected time of death less than three hours after NICU admission. Parents were excluded if they had mental health or language issues that might limit their integration and communication with the healthcare team.

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Depression reported by parents. | Survey completed by both parents one week after discharge.
  Use the Chinese version of the Hamilton Depression rating scale (HAMD) to evaluate depression among fathers. The Chinese version of the EPDS was used to assess depression among mothers.
  The HAMD includes 17 items with a 3 or 5-point Likert answer option scale with a total score of 78. The EPDS includes 10 items with a 4-point Likert answer option scale with a total score of 30. The higher scores means worse outcome.
satisfaction rate | Survey completed by both parents one week after discharge.
  Parent satisfaction was measured by the hospital standard parent satisfaction survey completed by both parents one week after discharge.The parent satisfaction instrument includes 20 items using a 5-point Likert answer option scale with a total score of 100.The higher scores means better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Children's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] Silverman WA. A hospice setting for humane neonatal death. Pediatrics. 1982 Feb;69(2):239. No abstract available. PMID 7058104
- [Background] Kim S, Savage TA, Hershberger PE, Kavanaugh K. End-of-Life Care in Neonatal Intensive Care Units from an Asian Perspective: An Integrative Review of the Research Literature. J Palliat Med. 2019 Jul;22(7):848-857. doi: 10.1089/jpm.2018.0304. Epub 2019 Jan 11. PMID 30632880
- [Result] Haug S, Dye A, Durrani S. End-of-Life Care for Neonates: Assessing and Addressing Pain and Distressing Symptoms. Front Pediatr. 2020 Sep 24;8:574180. doi: 10.3389/fped.2020.574180. eCollection 2020. PMID 33072678
- [Result] Dombrecht L, Beernaert K, Chambaere K, Cools F, Goossens L, Naulaers G, Cohen J, Deliens L; NICU consortium. End-of-life decisions in neonates and infants: a population-level mortality follow-back study. Arch Dis Child Fetal Neonatal Ed. 2022 May;107(3):340-341. doi: 10.1136/archdischild-2021-322108. Epub 2021 Jun 15. No abstract available. PMID 34131039
- [Result] Veldhuijzen van Zanten S, Ferretti E, MacLean G, Daboval T, Lauzon L, Reuvers E, Vadeboncoeur C. Medications to manage infant pain, distress and end-of-life symptoms in the immediate postpartum period. Expert Opin Pharmacother. 2022 Jan;23(1):43-48. doi: 10.1080/14656566.2021.1965574. Epub 2021 Aug 18. PMID 34384318
- [Result] Allen JD, Shukla R, Baker R, Slaven JE, Moody K. Improving Neonatal Intensive Care Unit Providers' Perceptions of Palliative Care through a Weekly Case-Based Discussion. Palliat Med Rep. 2021 Apr 16;2(1):93-100. doi: 10.1089/pmr.2020.0121. eCollection 2021. PMID 34223508
- [Result] Chen X, Li H, Song J, Sun P, Lin B, Zhao J, Yang C. The Resuscitation of Apparently Stillborn Neonates: A Peek Into the Practice in China. Front Pediatr. 2020 Jun 2;8:231. doi: 10.3389/fped.2020.00231. eCollection 2020. PMID 32582582
- [Result] Maurer DM, Raymond TJ, Davis BN. Depression: Screening and Diagnosis. Am Fam Physician. 2018 Oct 15;98(8):508-515. PMID 30277728
- [Result] Nixon N, Guo B, Garland A, Kaylor-Hughes C, Nixon E, Morriss R. The bi-factor structure of the 17-item Hamilton Depression Rating Scale in persistent major depression; dimensional measurement of outcome. PLoS One. 2020 Oct 26;15(10):e0241370. doi: 10.1371/journal.pone.0241370. eCollection 2020. PMID 33104761
- [Result] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Derived] Zhang R, Tang Q, Zhu LH, Peng XM, Zhang N, Xiong YE, Chen MH, Chen KL, Luo D, Li X, Latour JM. Testing a Family Supportive End of Life Care Intervention in a Chinese Neonatal Intensive Care Unit: A Quasi-experimental Study With a Non-randomized Controlled Trial Design. Front Pediatr. 2022 Jul 22;10:870382. doi: 10.3389/fped.2022.870382. eCollection 2022. PMID 35935359
- See also: World Health Organization. World Health Statistics 2021. Monitoring health for the SDGs. — https://apps.who.int/iris/bitstream/handle/10665/342703/9789240027053-eng.pdf
- See also: World Health Organization. Palliative Care. Key Facts. — https://www.who.int/news-room/fact-sheets/detail/palliative-care
- See also: National Institute for Health and Care Excellent (NICE). End of life care for infants, children and young people with life-limiting conditions: planning and management. NICE guideline — http://www.nice.org.uk/guidance/ng61